CLINICAL TRIAL: NCT01184742
Title: 6 Minute Push and 30 Second Sprint Tests Reliability and Relationship to Fitness, Participation, and Environmental Assessments
Brief Title: 6 Minute Push & 30 Second Sprint Tests Reliability & Relationship to Fitness, Participation, & Environmental Assessments
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Paralyzed Veterans of America (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Other Study IDs: TMP-MN-001
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2011-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the relationship between physical fitness and wheelchair mobility capacity and 1) participation; 2) self-reported environments barriers; and 3) self-reported avoidance of environmental features.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year post-injury
* able to self-propel a manual wheelchair
* spinal cord injury between C5 and T5

Exclusion Criteria:

* spinal cord injury above C5 or below T5
* spinal cord injury severity of AIS D
* unstable angina or myocardial infarction within the past month
* resting heart rate >120
* systolic blood pressure >180 mm Hg, or diastolic blood pressure >100 mm HG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of persons with spinal cord injury.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
6 Minute Push Test | Visit 3 and 4
30 Second Sprint Test | Visit 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States